CLINICAL TRIAL: NCT00236730
Title: Double-Blind Parallel Comparison of Three Doses of Topiramate and Placebo in Refractory Partial Epilepsy
Brief Title: A Study of the Efficacy and Safety of Topiramate in the Treatment of Patients With Difficult to Control Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005458
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Epilepsy; Epilepsies, Partial; Seizures
Keywords: topiramate; epilepsy; partial epilepsies; partial epilepsy; seizures; epileptic seizures; partial seizure disorder; brain diseases
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Seizures; Brain Diseases | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of topiramate as add-on therapy in patients with difficult to control partial onset seizures who are taking one or two standard anti-epileptic drugs.

DETAILED DESCRIPTION:
Epilepsy is characterized by seizures, which are abnormal electrical discharges in the brain that temporarily disrupt normal brain function. Seizures are classified as "generalized," originating in both sides of the brain simultaneously, or "partial-onset," starting in one area of the brain. Antiepilepsy medications, such as topiramate, are selected based on seizure type. This is a double-blind, placebo-controlled study that includes a baseline phase and a treatment phase. During the baseline phase (12 weeks duration), patients receive one or two of the following standard antiepileptic drugs (AEDs): phenytoin, carbamazepine, phenobarbital, or primidone. Patients who continue to have seizures during treatment with standard AEDs proceed into the double-blind treatment phase. Patients then receive placebo or topiramate at a dosage of 100-milligrams (mg) once daily, increasing to twice daily dosing at a maximum dose of 200 mg/day, 400 mg/day, or 600 mg/day or maximum tolerated dose (depending on treatment group), through Week 16 (total duration of double-blind phase), while continuing on their standard AED regimen. Assessments of effectiveness include the percent reduction in the average monthly seizure rate, percent of patients responding to treatment (having equal to or greater than 50% reduction in seizure rate), and, the patient's and investigator's global assessments of medication at end of study. Safety assessments include the incidence of adverse events throughout the study, clinical laboratory tests (hematology, serum chemistry, urinalysis), neurologic examinations, and vital sign measurements (blood pressure, pulse, temperature) weekly during the treatment phase. The study hypothesis is that topiramate, taken as add-on therapy to treatment with AEDs, will significantly reduce seizure frequency, compared with placebo, in patients with refractory partial epilepsy and is well-tolerated. Topiramate, 100 milligrams[mg] oral tablets. Dosage begins at 100-mg once daily and increases gradually to twice daily dosing at a maximum dose of 200, 400, or 600 mg/day, and continues through Week 16 (total duration).

ELIGIBILITY:
Inclusion Criteria:

* History of simple or complex partial epilepsy that has been documented or witnessed
* during a 12-week baseline phase, patient must have at least 12 partial seizures while maintaining therapeutic levels of antiepileptic drugs (AEDs)
* and have no more than one seizure-free interval of up to 3 weeks and none longer than 3 weeks
* good physical health.

Exclusion Criteria:

* Patients having solely generalized seizures or lacking documentation of partial epilepsy
* patients with generalized tonic-clonic seizures or other generalized epilepsies in the absence of an EEG consistent with partial epilepsy
* generalized seizures, which are defined by the EEG wave pattern
* seizures that lack an abnormal pulsation pattern on EEG
* females who are capable of having children

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 1988-06; Study Completion 1990-12 (Actual)

PRIMARY OUTCOMES:
Percent reduction in the average monthly seizure rate from baseline to end of treatment

SECONDARY OUTCOMES:
Percent of patients responding to treatment (>= 50% reduction in seizure rate from baseline to end of treatment); patient's and investigator's global assessments at end of study; incidence of adverse events throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Faught E, Wilder BJ, Ramsay RE, Reife RA, Kramer LD, Pledger GW, Karim RM. Topiramate placebo-controlled dose-ranging trial in refractory partial epilepsy using 200-, 400-, and 600-mg daily dosages. Topiramate YD Study Group. Neurology. 1996 Jun;46(6):1684-90. doi: 10.1212/wnl.46.6.1684. PMID 8649570
- See also: A study of the efficacy and safety of topiramate in the treatment of patients with difficult to control partial epilepsy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=645&filename=CR005458_CSR.pdf